CLINICAL TRIAL: NCT02905500
Title: Estimation Des années de Vie ajustées Sur l'incapacité à La réunion et Comparaison à la France métropolitaine et Aux Pays de la Zone Océan Indien
Brief Title: Estimation of Disability Adjusted Life Years in Reunion Island and Comparison to Metropolitan France and Other Countries in the Indian Ocean Zone
Acronym: AVIRON
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/CHU/AVIRON
Record Dates: First submitted 2016-09-12; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Quality-Adjusted Life Years; Epidemiology; Public Health
Keywords: Disability-Adjusted Life Years; Epidemiology; Public Health

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
AVIRON study aims at estimating the burden of various causes of death and morbidity in the Reunion Island population.

DETAILED DESCRIPTION:
The identification of health priorities on a given territory is a major field of the research in Public health. The World Health Organization leads since the 1990s the "Global Burden of Disease" study. This study has for objective to estimate the burden of various causes of death and morbidity in a given population. It defines a standardized measure allowing the comparisons between the various countries. The measure developed internationally is the Disability-adjusted life year (DALY).

For the Indian Ocean zone, the international study provides values of DALYs for Madagascar, Seychelles and Mauritius. The estimation of DALYs for Reunion Island are based on data of mainland France and does not take into account specificities from Reunion Island. To better define Public health priorities, it seems essential to decline this measure at the regional level.

ELIGIBILITY:
Inclusion Criteria:

* The whole population of Reunion Island

Exclusion Criteria:

* People not living in Reunion Island

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Resident of Reunion Island
Sampling Method: Non-Probability Sample
Enrollment: 800000 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of years of life lost or lived with disabilities | 3 years
Prevalence of years of life lost or lived with disabilities | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Universitaire de La Réunion, Saint-Pierre, France